CLINICAL TRIAL: NCT00351234
Title: Correlation Between Carnitine Deficiency and Hypoglycemic Events in Type I Diabetes; Effects of Carnitine Supplementation on Hypoglycemic Events in Type I Diabetes
Brief Title: Carnitine Levels and Carnitine Supplementation in Type I Diabetes
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Leadiant Biosciences, Inc. (Industry); Minimed Pharmaceuticals (Industry); Pharmacia/Upjohn Career Development Award (Unknown)
Responsible Party: L. Kurt Midyett, MD, Assistant Professor, Children's Mercy Hospital
Other Study IDs: 000003020
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus, Type I; Hypoglycemia
Keywords: Diabetes Mellitus Type I,; Hypoglycemia,; Carnitine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Carnitine; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Carnitine (drug) — Oral L-carnitine will be obtained from Sigma Tau Pharmaceuticals. Supplementation will be initiated at 50mg/kg body weight and increased to 100mg/kg body weight after one week.

SUMMARY:
The purpose of this study is to determine whether type I diabetics with carnitine deficiency exhibit increased numbers of hypoglycemic (low blood sugars) events and if unrecognized hypoglycemia occurs during continuous 72-hour glucose monitoring. If they are determined to have unrecognized hypoglycemia, then oral carnitine supplementation will be given to those subjects and they will be reassessed for the number of hypoglycemic events in a 72-hour glucose monitoring.

DETAILED DESCRIPTION:
Hypoglycemia is a clinical marker of carnitine deficiency. Thus carnitine may compound the risk of hypoglycemia for children on insulin therapy. Currently, one of the limitations in the management of diabetes is hypoglycemia. The problem of hypoglycemia is of even greater significance in the pediatric population because children have smaller glycogen stores.

In this study, we will determine if there is a group of children with increased frequency of hypoglycemia and carnitine deficiency. If there is a correlation from the initial 200 children, we will compare two groups of type I diabetic children between the ages of 7 to 21 years. We will take 20 children with the highest carnitine levels (found in a previous study) and 20 children with the lowest carnitine levels and perform continuous glucose monitoring for a 72-hour period. Those who have at least one episode of hypoglycemia will be asked to undergo repeat testing, after a 2-week period of oral carnitine supplementation. Supplementation will start at 50 mg/kg body weight for the first week and then increase to 100 mg/kg body weight the second week. Laboratory studies obtained at baseline include Hemoglobin A1c, carnitine panel, and lipid panel. These will be repeated prior to the second continuous glucose monitoring. Insulin doses will not be changed between glucose monitoring sessions. A comparison will be made between individuals with hypoglycemia, to see if the number of hypoglycemic events has decreased.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type I for greater than 2 years between the ages of 7 and 21
* currently on insulin replacement therapy

Exclusion Criteria:

* Patients with newly diagnosed Type I diabetes
* Patients already taking L-carnitine
* Patients who come to clinic without glucose monitors
* Patients with known seizure disorders not including hypoglycemic seizures
* Patients on metformin
* Patients with compromised renal function.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Children (male or female), between the ages of 7 and 21,
  2. who have had a diagnosis of Type 1 diabetes mellitus for at least two years and
  3. are currently on insulin replacement therapy.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2004-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To see if there is a correlation between carnitine levels and number of hypoglycemic events. | one year
To see if carnitine values in a control population are significantly different than our study group. | one year
To see if the number of hypoglycemic events decreases with treatment of carnitine on type I diabetic patients. The measurements will be taken after the second 72-hour continuous glucose monitoring. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Midyett, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Rebouche CJ, Paulson DJ. Carnitine metabolism and function in humans. Annu Rev Nutr. 1986;6:41-66. doi: 10.1146/annurev.nu.06.070186.000353. PMID 3524622
- [Background] Frohlich J, Seccombe DW, Hahn P, Dodek P, Hynie I. Effect of fasting on free and esterified carnitine levels in human serum and urine: correlation with serum levels of free fatty acids and beta-hydroxybutyrate. Metabolism. 1978 May;27(5):555-61. doi: 10.1016/0026-0495(78)90022-7. PMID 642827
- [Background] Hoppel CL, Genuth SM. Urinary excretion of acetylcarnitine during human diabetic and fasting ketosis. Am J Physiol. 1982 Aug;243(2):E168-72. doi: 10.1152/ajpendo.1982.243.2.E168. PMID 6810706
- [Background] Bohles H, Evangeliou A, Bervoets K, Eckert I, Sewell A. Carnitine esters in metabolic disease. Eur J Pediatr. 1994;153(7 Suppl 1):S57-61. doi: 10.1007/BF02138779. No abstract available. PMID 7957388
- [Background] Soltesz G, Melegh B, Sandor A. The relationship between carnitine and ketone body levels in diabetic children. Acta Paediatr Scand. 1983 Jul;72(4):511-5. doi: 10.1111/j.1651-2227.1983.tb09762.x. PMID 6353846
- [Background] Winter SC, Simon M, Zorn EM, Szabo-Aczel S, Vance WH, O'Hara T, Higashi L. Relative carnitine insufficiency in children with type I diabetes mellitus. Am J Dis Child. 1989 Nov;143(11):1337-9. doi: 10.1001/archpedi.1989.02150230095030. PMID 2816861
- [Background] Pons R, De Vivo DC. Primary and secondary carnitine deficiency syndromes. J Child Neurol. 1995 Nov;10 Suppl 2:S8-24. PMID 8576570
- [Background] Stanley CA. New genetic defects in mitochondrial fatty acid oxidation and carnitine deficiency. Adv Pediatr. 1987;34:59-88. PMID 3318304
- [Background] O'Donnell J, Finer NN, Rich W, Barshop BA, Barrington KJ. Role of L-carnitine in apnea of prematurity: a randomized, controlled trial. Pediatrics. 2002 Apr;109(4):622-6. doi: 10.1542/peds.109.4.622. PMID 11927706
- [Background] Maebashi M, Kawamura N, Sato M, Imamura A, Yoshinaga K. Lipid-lowering effect of carnitine in patients with type-IV hyperlipoproteinaemia. Lancet. 1978 Oct 14;2(8094):805-7. doi: 10.1016/s0140-6736(78)92587-4. PMID 81361